CLINICAL TRIAL: NCT05036278
Title: A Multicenter, Prospective, Open-label, Clinical Study to Assess the Effect of Using a New Risk Score Approach to Select the Most Appropriate Prophylaxis Regimen for Reaching a Favorable Outcome, When Hemophilia A Patients Switch From Standard Half-life Products to Damoctocog Alfa Pegol (Jivi)
Brief Title: Prophylaxis Regimen for Hemophilia A Patients
Acronym: PREDICT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21924; 2021-006191-16 (EudraCT Number)
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A; Prophylaxis of Bleeding
MeSH Terms: conditions — Hemophilia A | interventions — Polyethylene Glycols; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Damoctocog alfa-pegol prophylaxis regimens (Experimental): Prophylaxis regimens: All participants will begin with prophylaxis 2x/week (40 IU/kg/dose (recommended maximum dose 6,000 IU)) Participants with a high risk score (> 4) continue on prophylaxis 2x/week (40 IU/kg/dose). Participants with a medium risk score (2 to 4) will switch after 4 weeks to prophylaxis Q5D (50 IU/kg/dose). Participants with a low risk score (< 2) will switch after 4 weeks to prophylaxis Q5D (50 IU/kg/dose) and then after 4 weeks to a less frequent (e.g. Q7D) regimen (60 IU/kg/dose).
  Interventions: Biological: Damoctocog alfa-pegol is a recombinant B-domain deleted human coagulation FVIII variant site specifically conjugated with a 60 kDa, branched (30 kDa each) polyethylene glycol (PEG).

INTERVENTIONS:
Biological: Damoctocog alfa-pegol is a recombinant B-domain deleted human coagulation FVIII variant site specifically conjugated with a 60 kDa, branched (30 kDa each) polyethylene glycol (PEG). — Dosage Levels:
  * 40 IU/kg/dose two times per week
  * 50 IU/kg/dose every 5 days
  * 60 IU/kg/dose, Less frequent dosing (e.g. every 7 days), the total recommended maximum dose/infusion is 6000 IU.
  Other Names: Jivi, BAY94-9027

SUMMARY:
Researchers are looking for a better way to treat people who have hemophilia A. Hemophilia A is a genetic bleeding disorder that is caused by the lack of a protein in the blood called "clotting factor 8" (FVIII). FVIII is naturally found in the blood where it causes the blood to clump together to help prevent and stop bleeding. People with lower levels of FVIII or with FVIII that does not work properly may bleed for a long time from minor wounds, have painful bleeding into joints, or have internal bleeding.

The study treatment, Jivi (also called damoctocog alfa pegol), is already available for doctors to prescribe to people with hemophilia A to treat and prevent bleeding. It works by replacing the missing FVIII, or the FVIII that does not work properly.

People with hemophilia A need frequent injections of FVIII products into the vein. So called standard half-life (SHL) products need to be given 2 to 4 times a week for the prevention of bleeding. In recent years, new products like Jivi called extended half-life (EHL) products have become available. These products last longer in the body so that they require to be given less often with injections every 3-5 days. Thus, these treatments may be easier and more comfortable to stick to in daily life. There is no general plan concerning the best amount of treatment and the frequency of injections for the prevention of bleeding, since the severity may be different and individual risk factors have to be considered. Doctors often decide on a treatment plan based on their experience.

The main purpose of this study is to learn how well a new scoring approach works to select a treatment plan for the prevention of bleeding in people with hemophilia A who switch their treatment from SHL products to Jivi. Different types of information are used to calculate the risk score like bleeding history, certain biological factors, and physical activity of the participant.

All participants will receive Jivi for 6 months.

In the first four weeks, all participants will receive Jivi 2 times a week at a dose level of 40 IU per kilogram body weight (also known as 40 IU/kg/dose, recommended maximum dose is 6,000 IU). Then, based on their risk score, each participant will be assigned to one of three treatment plans:

* participants with a high risk remain on Jivi administration 2 times a week at 40 IU/kg/dose
* participants with a medium risk will switch to Jivi administration every 5 days at 50 IU/kg/dose
* participants with a low risk will switch to Jivi administration every 5 days at 50 IU/kg/dose and after 4 weeks to a less frequent administration (e.g., every 7 days) at 60 IU/kg/dose To check how well the new scoring approach works for choosing the right treatment plan, researchers will look at how many participants have a favourable outcome.

This means that the participant has either fewer bleeding events vs. the pre-study treatment and takes Jivi less often or as often as the previous SHL treatment but with fewer bleeding events, or that the participant has a comparable number of bleeding events but needs to take Jivi less often than the previous treatment. Each participant will be in the study for approximately 7.5 months. During this time, 4 visits to the study site and 3 phone calls are planned. During the study, the doctors and their study team will: • do physical examinations • take blood samples • ask the participants questions about how they are feeling and what adverse events they are having. In addition, participants or their guardians are required to write down the dates of Jivi treatments and bleeding events in an electronic diary and to fill in different questionnaires on their quality of life, health status, work/ school productivity, pain, and treatment satisfaction. In addition, participants are expected to keep appointments for visits and to adhere to the assigned treatment regimen.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 12 years of age inclusive, at the time of signing the informed consent/assent.
* Previously treated patients (≥ 150 EDs) with congenital hemophilia A.
* Prophylaxis with any SHL FVIII product with a stable frequency for at least 6 consecutive months within the last 12 months prior to screening before entering the study and documented in medical records. Stable frequency is defined as a minimum 18 weeks of treatment in a 6 (consecutive) calendar month period in the 12 months prior to screening. Patients can be on any non-Jivi EHL between the 6-month stable SHL prophylaxis period and start of study treatment.
* Documented bleeding rate (ABR) while on stable frequency SHL prophylaxis for at least 6 consecutive months within the last 12 months prior to screening.
* No current evidence (≥ 0.6 BU/mL) of FVIII inhibitors. If a participant has had a positive inhibitor titer in the past (≥ 0.6 BU/mL on two occasions) but has been tolerized for at least 1 year since the last positive titer with at least 1 negative inhibitor assay test during that period, they can be enrolled. If a participant has had a positive inhibitor titer in the past (≥ 0.6 BU/mL) but did not require tolerization and has had at least 1 negative inhibitor assay test during a minimum period of at least 1 year since the last positive titer, they can be enrolled.
* If they are human immunodeficiency virus (HIV) positive, cluster of differentiation 4 (CD4+) lymphocyte count should be > 200/mm^3 within 1 year before entering the study and documented in medical records. -
* Participants who are willing to complete an electronic diary (eDiary).
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* For adolescent participants (≥ 12 to < 18 years), a legal guardian must be available to help the study-site personnel ensure follow-up; accompany the participant to the study site on each assessment day according to the Schedule of Activities (SoA) (e.g. able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures); consistently and consecutively be available to provide information on the participant using the PROs during the scheduled study visits; accurately and reliably dispense study intervention as directed.
* For adolescent participants, a legal guardian must be able to accurately maintain the child's take-home record, including items of general health.

Exclusion Criteria:

* Any other inherited or acquired bleeding disorder in addition to hemophilia A. Note: von Willebrand disease should be diagnosed per local clinical practice. Participants with a diagnosis of von Willebrand disease in medical records or diagnosed at the time of screening will be excluded.
* Platelet count < 100,000/mm^3
* Evidence of inhibitor to FVIII (≥ 0.6 BU/mL) within the last 1 year
* The participant is currently participating in another investigational drug study or has participated in a clinical study involving an investigational drug or device within 30 days of signing informed consent.
* The participant has a planned major surgery.
* Documentation of missing risk score parameters other than physical activity .
* Known hypersensitivity to the drug substance, excipients, or mouse or hamster protein.
* Any other significant medical condition that the investigator feels would be a risk to the participant or would impede the study.
* Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site).
* Otherwise vulnerable participants (e.g. participants who are in custody by order of an authority).
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures (i.e. eDiary completion, clinic visits, phone updates), restrictions, and requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Dr. Akshat Jain - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University Children's Hospital - Hematology / Oncology, Loma Linda, California
  - Luskin Orthopaedic Institute for Children, Los Angeles, California
  - University of Colorado | Renal Research Office, Aurora, Colorado
  - UHealth - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Aflac Cancer and Blood Disorders Center - Egleston Hospital, Atlanta, Georgia
  - Wellstar MCG Health Medical Center - Gynecology, Augusta, Georgia
  - Rush University Medical Center - Oncology, Chicago, Illinois
  - Stead Family Children's Hospital - Hematology / Oncology, Iowa City, Iowa
  - M Health Fairview Masonic Cancer Clinic - Clinics and Surgery Center, Minneapolis, Minnesota
  - Rutgers Robert Wood Johnson Medical School - OBGYN, New Brunswick, New Jersey
  - Gulf States Hemophilia & Thrombophilia Center- Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 study centers in the US between 28 July 2022 (first particpant first visit) and 12 September 2024 (last participant last visit).
Pre-assignment Details: A total of 21 participants were enrolled. 21 participants were assigned to treatment.
Groups:
- Overall Study: 2x/week (40 IU/kg/dose) with Jivi for 4 weeks, continued according to assigned prophylaxis regimen.
Period: Overall Study
Arm/Group | Overall Study
Started (21) | 21
Completed (19) | 19
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: 2x/week (40 IU/kg/dose) with Jivi for 4 weeks, continued according to assigned prophylaxis regimen.
Arm/Group | Overall
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 3
  Adults (18-64 years) | 17
  From 65-84 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Number of Participants With Favorable Outcome on the Score-assigned Prophylaxis Regimen
Description: Overall number of participants with favorable outcomes after prophylaxis regimen assignment by a risk score, based on a participant's baseline phenotypic and biologic variables, when switching from a standard half-life (SHL) product to Jivi.
Time Frame: up to 6 months
Population: all patients enrolled, followed for at least 4 months and not having switched from the prophylaxis regimen, determined by the risk-score; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Number; unit: participants
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 17
participants | 12

2. Secondary Outcome: Annualized Bleeding Rate (ABR) (Total, Joint, Spontaneous)
Description: To assess the efficacy of Jivi
Time Frame: up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 17
bleeds per year
  total bleeds | 4.172 (5.516)
  joint bleeds | 2.800 (4.160)
  spontaneous bleeds | 1.788 (3.968)

3. Secondary Outcome: Change in Total ABR From Pre-study
Description: To assess the efficacy of Jivi compared to a previous SHL treatment.
Time Frame: up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 17
bleeds per year | -8.005 (15.242)

4. Secondary Outcome: Change in the Frequency of Pre-study SHL Teratment to the Frequency of Jivi Administration (Infusions/Month)
Description: To assess the frequency of Jivi administration.
Time Frame: up to 6 months
Population: all patients enrolled, followed for at least 4 months; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Mean (Standard Deviation); unit: infusions per month
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 17
infusions per month | -6.876 (4.7557)

5. Secondary Outcome: Occurrence of Participants With 0 and ≤ 1 Spontaneous Bleeds
Description: To assess the proportion of participants with 0 and ≤ 1 spontaneous bleeds.
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Number; unit: participants
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 19
participants
  0 spontaneous bleed | 13
  <=1 spontaneous bleeds | 13

6. Secondary Outcome: Change in Haemophilia Quality of Life Questionnaire (Haem-A-QoL or Haemo-QoL)
Description: To assess participant quality of life (QoL) and physical activity, as measured by the Patient Reported Outcomes (PROs) Hemophilia A-specific quality of life and Hemophilia-specific quality of life. This includes 41 items covering 6 domains: Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact, and Treatment Concerns. The Haemo-QoL Short Form contains 35 items covering 9 domains: Physical Health, View of Yourself, Family, Friends, Others, Sports, Dealing, and Treatment. A higher score on the questionnaire represents greater impairment, and a negative change from baseline represents improvement. The percentage score is sum of item scores divided by the possible range. Individual item scores range from 1 to 5.
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months, only 10 participants completed this patient-reported outcome; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Mean (Standard Deviation); unit: Percentage of scores on a scale
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 19
Percentage of scores on a scale
  Visit 2 (Baseline): number analyzed (Participants) | 14
  Visit 2 (Baseline) | 31.5 (16.38)
  Change from baseline at visit 6: number analyzed (Participants) | 10
  Change from baseline at visit 6 | -4.7 (11.7)

7. Secondary Outcome: Patient's Global Impression of Change (PGI-C)
Description: To assess participant quality of life (QoL) and physical activity, as measured by Patient-Reported Outcomes (PROs).
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months, only 9 participants completed this patient-reported outcome; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Count of Participants; unit: Participants
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 9
Participants
  status minimally improved | 1
  status minimally worse | 1
  status much improved | 2
  status not changed | 4
  status very much improved | 1

8. Secondary Outcome: EuroQoL 5 Dimensions (EQ-5D-5L) Questionnaire
Description: To assess participant quality of life (QoL) and physical activity, as measured by Patient-Reported Outcomes (PROs). Change to baseline means changes between Visit 2 and Visit 6
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months, only 11 participants completed this patient-reported outcome; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Count of Participants; unit: Participants
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 11
Participants
  walking: improved, less impaired | 1
  walking: no change | 5
  walking: worsened, more impaired | 5
  self-care: improved, less impaired | 1
  self-care: no change | 10
  self-care: worsened, more impaired | 0
  usual activity: improved, less impaired | 0
  usual activity: no change | 11
  usual activity: worsened, more impaired | 0
  pain or discomfort: improved, less impaired | 0
  pain or discomfort: no change | 9
  pain or discomfort: worsened, more impaired | 2
  anxious or depressed: improved, less impaired | 2
  anxious or depressed: no change | 6
  anxious or depressed: worsened, more impaired | 3

9. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: To assess participant quality of life (QoL) and physical activity, as measured by Patient-Reported Outcomes (PROs). Score ranges from 10 (lowest satisfaction) to 100 (greatest satisfaction).
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months, only 5 participants completed this patient-reported outcome; This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 5
Percentage
  Visit 2 (baseline) | 37.9 (7.44)
  Change from baseline at visit 6 | -1.8 (6.42)

10. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire Scores
Description: Work Productivity and Activity Impairment Questionnaire scores for hemophilia effect over the last 7 days on productivity or ability at work, at school, and in regular daily activities. It ranges from 0% to 100%, where higher scores indicate greater work impairment and less productivity.
  To assess participant quality of life (QoL) and physical activity, as measured by Patient Reported Outcomes (PROs). Baseline = Visit 2, Change from Baseline = Visit 6
Time Frame: up to 6 months
Population: All participants enrolled and followed for at least 4 months, participants' number completing this patient-reported outcome varied depending on parameter;This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 19
Percentage
  Percent Work Time Missed (baseline) 7 participants: number analyzed (Participants) | 7
  Percent Work Time Missed (baseline) 7 participants | 1.8 (4.64)
  Percent Work Time Missed (change from baseline) 4 participants: number analyzed (Participants) | 4
  Percent Work Time Missed (change from baseline) 4 participants | 19.4 (24.21)
  Percent Working Impairment (baseline) 6 participants: number analyzed (Participants) | 6
  Percent Working Impairment (baseline) 6 participants | 26.7 (22.51)
  Percent Working Impairment (change from baseline) 3 participants: number analyzed (Participants) | 3
  Percent Working Impairment (change from baseline) 3 participants | 10.0 (20.00)
  Percent Class Time Missed (baseline) 4 participants: number analyzed (Participants) | 4
  Percent Class Time Missed (baseline) 4 participants | 5.0 (10.00)
  Percent Class Time Missed (change from baseline) 2 participants: number analyzed (Participants) | 2
  Percent Class Time Missed (change from baseline) 2 participants | 1.4 (1.96)
  Percent Class Attending Impairment (baseline) 4 participants: number analyzed (Participants) | 4
  Percent Class Attending Impairment (baseline) 4 participants | 15.0 (19.15)
  Percent Class Attending Impairment (change) 2 participants: number analyzed (Participants) | 2
  Percent Class Attending Impairment (change) 2 participants | 0 (28.28)
  Percent Daily Activities Impairment (baseline) 12 participants: number analyzed (Participants) | 12
  Percent Daily Activities Impairment (baseline) 12 participants | 33.3 (29.34)

11. Secondary Outcome: Number of Target Joints and Change in Target Joint Status From Baseline
Description: To assess target joint status, per modified International Society on Thrombosis and Haemostasis (ISTH) guidelines
Time Frame: up to 6 months
Population: as for outcome 5
Measure: Number; unit: Joints
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
Number analyzed (Participants) | 19
Joints
  zero (baseline) | 8
  one (baseline) | 4
  two (baseline) | 2
  three (baseline) | 3
  four (baseline) | 2
  minus four (change from baseline) | 1
  minus three (change from baseline) | 4
  minus two (change from baseline) | 2
  minus one (change from baseline) | 4
  zero (change from baseline) | 8

ADVERSE EVENTS:
Time Frame: All Adverse events were collected from the first study intervention up to 14 days after the end of study intervention, an average of 7 months.
Description: Treatment Emergent AEs for Safety Population, i.e. all participants who have received at least one study intervention.
  This analysis included only one single arm. Within this single arm, each participant was assigned a prophylaxis regimen according to a risk score, based on a participant's phenotypic and biologic variables.
Arm/Group | Damoctocog Alfa-pegol Prophylaxis Regimens
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Damoctocog Alfa-pegol Prophylaxis Regimens (N=21)
Haemorrhage (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Damoctocog Alfa-pegol Prophylaxis Regimens (N=21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigative Site/Institution/ Principal Investigator have the right to publish the results of their activities only in accordance with the agreement and if they do not constitute a violation of the Confidential Information. They agree to submit any proposed publication to Sponsor for review. The sponsor has the right to require removal of specifically identified Confidential Information and/or to delay the proposed Publication for an additional 30-60 days.

DOCUMENTS (2):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT05036278/Prot_004.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT05036278/SAP_005.pdf